CLINICAL TRIAL: NCT00046943
Title: A Phase III Extension Study to Evaluate the Safety of 10 mg Atrasentan in Men With Hormone-Refractory Prostate Cancer
Brief Title: Atrasentan in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000257127; ABBOTT-M00-258; UCLA-0202002; NCI-G02-2110
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2003-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Atrasentan

INTERVENTIONS:
Drug: atrasentan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase III trial to determine the effectiveness of atrasentan in treating patients who have prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of atrasentan in patients with hormone-refractory prostate cancer.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral atrasentan once daily for 3 years in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month and then every 3 months for 2 years.

PROJECTED ACCRUAL: Approximately 1,400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hormone-refractory prostate cancer
* Completed protocol ABBOTT-M00-211 or ABBOTT-M00-244 within the past 30 days

  * Disease progression OR
  * Active in trial when double-blind treatment period ended

PATIENT CHARACTERISTICS:

Age

* 19 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm3
* Absolute neutrophil count greater than 1,000/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9 g/dL

Hepatic

* Bilirubin less than 1.5 mg/dL
* AST and ALT no greater than 1.5 times upper limit of normal

Renal

* Creatinine clearance at least 40 mL/min

Cardiovascular

* No New York Heart Association class II-IV heart disease

Pulmonary

* No significant pulmonary disease requiring chronic or pulse steroid therapy within the past 3 months

Other

* Fertile patients must use 2 effective methods of contraception (1 must be barrier contraception) during and for 8 weeks after study
* No reason that would preclude study
* No significant comorbid condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since other prior cytotoxic chemotherapy
* No other concurrent cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radionuclides
* No concurrent radionuclides

Surgery

* Not specified

Other

* At least 4 weeks since prior investigational agents
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent participation in another investigational study

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Gordon, MD, PhD — Abbott
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States